CLINICAL TRIAL: NCT03301103
Title: PTM202 and Modulation of Host Resistance to Diarrheagenic Escherichia Coli in a Randomized, Double-blind, Placebo Controlled Study in Healthy Human Subjects
Brief Title: PTM202 and Modulation of Host Resistance to Diarrheagenic E. Coli
Acronym: APA12/PANTER
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NIZO Food Research (Other)
Collaborators: PanTheryx, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NL62453.028.17
Record Dates: First submitted 2017-09-15; First posted 2017-10-04 (Actual); Last update posted 2018-07-18 (Actual); Status verified 2018-07

CONDITIONS: Traveler's Diarrhea
Keywords: Nutrition; Gastroenteritis; Traveler's diarrhea; E. coli
MeSH Terms: conditions — Gastroenteritis; Escherichia coli Infections

STUDY DESIGN:
Intervention Model Description: The APA12/PANTER study is a randomized, double-blind, placebo-controlled, parallel intervention study of 3 weeks in 72 healthy adults. Subjects will be orally infected with a live, but attenuated, diarrheagenic E. coli (strain E1392-75-2A; collection NIZO food research; dose 1E10 CFU (at study day 14). At study day 14, 15 and 16 subjects will receive either placebo or PTM202, a dietary formula containing dried bovine colostrum and dried whole egg.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: All researchers of the project team will be kept blind to assignment of treatment, and so will be the study subjects.The placebo will be matched in appearance and flavour to PTM202.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Placebo (Placebo Comparator): The placebo will consist of low-lactose isonitrogenous soy product, and will be matched in appearance and flavour to PTM202.
  After an overnight fast, subjects will be orally infected with a live, but attenuated, diarrheagenic E. coli (strain E1392-75-2A; collection NIZO food research; dose 1E10 CFU (at study day 14).
  Interventions: Biological: E. coli strain E1392-75-2A
- PTM202 (Experimental): PTM202 is a dry powder for reconstitution, comprised of a proprietary mixture of dried bovine colostrum and dried whole egg.
  After an overnight fast, subjects will be orally infected with a live, but attenuated, diarrheagenic E. coli (strain E1392-75-2A; collection NIZO food research; dose 1E10 CFU (at study day 14).
  Interventions: Biological: E. coli strain E1392-75-2A; Device: PTM202

INTERVENTIONS:
Biological: E. coli strain E1392-75-2A — After an overnight fast, subjects will be orally infected with a live, but attenuated, diarrheagenic E. coli (strain E1392-75-2A; collection NIZO food research; dose 1E10 CFU (at study day 14).
Device: PTM202 — PTM202 is a dietary formula containing a proprietary mixture of dried bovine colostrum and dried whole egg.
  Arms: PTM202

SUMMARY:
The APA12/PANTER study is a parallel 3-weeks intervention study. Subjects will be randomly assigned to one of two treatment groups; placebo or PTM202 (n=36 per group). After an overnight fast, subjects will be orally infected with a live, but attenuated, diarrheagenic E. coli at study day 14. At various time points before and after diarrheagenic E. coli challenge an online diary will be kept to record information on stool consistency, frequency and severity of symptoms and stool samples will be collected to determine total fecal wet weight and percentage of fecal wet weight.

DETAILED DESCRIPTION:
The APA12/PANTER study is a randomized, double-blind, placebo-controlled, parallel intervention study of 3 weeks in 72 healthy adults. The study will include 2 arms; PTM202 and placebo. Subjects will be instructed to maintain their usual pattern of physical activity and their habitual food intake, but to standardize their dietary calcium intake. After an overnight fast, subjects will be orally infected with a live, but attenuated, diarrheagenic E. coli (strain E1392-75-2A; collection NIZO food research; dose 1E10 CFU (at study day 14).

At study day 14, 15 and 16 subjects will receive either placebo or PTM202, a dietary formula containing dried bovine colostrum and dried whole egg.

Before and after the diarrheagenic E. coli challenge an online diary will be kept to record information on stool consistency, frequency, severity of symptoms and mediation intake. At various time points before and after diarrheagenic E. coli challenge stool samples will be collected. The main study parameters are Stool consistency (Bristol Stool Scale reported by the subjects in the online diary, and Percentage of fecal wet weight (% determined by freeze-drying).

Secondary study parameters are: Stool frequency (Stools per day reported by the subjects in the online diary), Total fecal wet weight (fecal weight in g/day), and the incidence and severity of Gastro-intestinal symptoms (Gastro-intestinal Symptom Rating Scale reported by the subjects in the online diary).

ELIGIBILITY:
Inclusion Criteria:

1. Male;
2. Age between 18 and 55 years;
3. BMI ≥18 and ≤27 kg/m2;
4. Healthy as assessed by the NIZO food research medical questionnaire.
5. Ability to follow verbal and written instructions;
6. Availability of internet connection;
7. Signed informed consent;
8. Willing to accept disclosure of the financial benefit of participation in the study to the authorities concerned;
9. Willing to accept use of all encoded data, including publication, and the confidential use and storage of all data for at least 15 years;
10. Willing to comply with study procedures, including collection of stool samples;
11. Willingness to abstain from high calcium containing products;
12. Willingness to abstain from alcoholic beverages three days before, during and for four days after diarrheagenic E. coli challenge;
13. Willingness to abstain from antibiotics, norit, laxatives, nonsteroidal anti-inflammatory drugs (OTC), opiates, antacids, proton pump inhibitors, and antimotility agents (e.g., loperamide) on the three days before, during and for four days after diarrheagenic E. coli challenge.
14. Willingness to abstain from probiotics three days before, during and for four days after diarrheagenic E. coli challenge;
15. Willingness to give up blood donation starting 1 month prior to study start and during the entire study;

Exclusion Criteria:

1. Any confirmed or suspected immunosuppressive or immunodeficient condition including human immunodeficiency virus infection (HIV);
2. Disease of the GI tract, liver, bile bladder, kidney, thyroid gland (self-reported);
3. Diarrheagenic E. coli strain (as used in the study) detected in fecal sample at screening;
4. Evidence of current excessive alcohol consumption or non-therapeutic drug (ab)use);
5. High titer serum antibodies against CFA-II diarrheagenic E. coli strain (as used in the study) at screening;
6. History of microbiologically confirmed ETEC or cholera infection in last 3 years;
7. Known allergy to the following antibiotics: ciprofloxacin, trimethoprim-sulfamethoxazole, and penicillins;
8. Known allergy to soy, milk- and/or egg;
9. Mental status that is incompatible with the proper conduct of the study;
10. Occupation involving handling of ETEC or Vibrio cholerae currently, or in the past 3 years;
11. Reported average stool frequency of <1 or >3 per day;
12. Symptoms consistent with Travelers' Diarrhea concurrent with travel to countries where ETEC infection is endemic (most of the developing world) within 3 years prior to dosing, OR planned travel to endemic countries during the length of the study;
13. Use of antibiotics, norit, laxatives (up till 6 months prior to inclusion), cholesterol lowering agents, antacids, proton pump inhibitors and immune suppressive agents (up till 3 months prior to inclusion);
14. Vaccination for or ingestion of ETEC, cholera, or E coli heat labile toxin within 3 years prior to inclusion;
15. Vegans.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Gender identity is self-reported by the subjects through a questionnaire.
Enrollment: 72 (Actual)
Dates: Start 2017-12-07 (Actual); Primary Completion 2018-01-23 (Actual); Study Completion 2018-03-16 (Actual)

PRIMARY OUTCOMES:
Stool consistency | Before challenge (Day 11-13), After challenge (Day 14-18)
  Change in stool consistency score (questionnaire) before and after E. coli challenge
Relative fecal wet weight | Before challenge (Day 11-13), After challenge (Day 14-18)
  Change in relative fecal wet weight (freeze-drying) before and after E. coli challenge

SECONDARY OUTCOMES:
Stool frequency | Before challenge (Day 11-13), After challenge (Day 14-18)
  Change in stool frequency (questionnaire) before and after E. coli challenge
Total fecal wet weight | Before challenge (Day 11-13), After challenge (Day 14-18)
  Change in total fecal wet weight (wet weight measurement) before and after E. coli challenge
Gastro-intestinal symptoms | Before challenge (Day 11-13), After challenge (Day 14-18)
  Change in gastro-intestinal symptoms (questionnaire) before and after E. coli challenge

CONTACTS AND LOCATIONS:
Overall Officials: Van Schaik, Study Director — NIZO Food Research
Locations (1):
- NIZO, Ede, Gelderland, Netherlands

IPD SHARING:
Plan to Share IPD: No